CLINICAL TRIAL: NCT06910189
Title: Use of Fish Skin Graft (FSG) to Improve Wound Healing and Expedite Discharge at a County Safety-net Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jonah Stulberg, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-24-1100
Record Dates: First submitted 2025-03-27; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Surgical Wound
Keywords: Fish Skin Graft (FSG); Kerecis
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients and nursing staff will be blinded to the patient's study arm. The operative physician will not be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fish Skin Graft arm and Vacuum-Assisted Closure (Experimental)
  Interventions: Device: Fish Skin Graft (FSG); Device: Wound Vacuum-Assisted Closure (VAC)
- Vacuum-Assisted Closure only (Active Comparator)
  Interventions: Device: Wound Vacuum-Assisted Closure (VAC)

INTERVENTIONS:
Device: Fish Skin Graft (FSG) — FSG will be applied to the wound bed, followed by a wound VAC at the time of surgical debridement
  Arms: Fish Skin Graft arm and Vacuum-Assisted Closure
Device: Wound Vacuum-Assisted Closure (VAC) — Participants will have a wound VAC applied to their wound bed at the time of surgical debridement.

SUMMARY:
The purpose of this study is to estimate the effect of FSG (Kerecis) on hospital length of stay among adult patients with surgical wounds of at least 40cm2 requiring surgical debridement

ELIGIBILITY:
Inclusion Criteria:

* Has wound greater than or equal to 40cm2 requiring surgical debridement
* Agreeable to follow up period of up to 1 year

Exclusion Criteria:

* Patients with wounds that do not require surgical debridement.
* Patients with a known allergy or other sensitivity to fish material
* Patients who are deemed unlikely to follow up (e.g., patients who live out of state).
* Patients in police custody/incarcerated.
* Patients unable to communicate in either Spanish or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | from time of admission to time of discharge (about 3 days from date of surgery)

SECONDARY OUTCOMES:
Number of participants that have recurrent surgical site infection | Upto 1 year after surgery
Number of participants that require reoperation | Upto 1 year after surgery
Time to total wound healing | From end of surgery to upto 1 year after surgery
Number of participants that need skin graft | Upto 1 year after surgery
time from original surgery with placement of wound vac until the patient gets a skin graft | upto 1 year after surgery
time to return to work | From discharge (about 3 days from date of surgery) upto 1 year after surgery
Number of participants that need wound vac after discharge | At discharge (about 3 days from date of surgery)
Inpatient hospital costs | At discharge (about 3 days from date of surgery)
financial toxicity experienced by patients as assessed by the COST - FACIT survey | 3 months after discharge
  This is a 12 item questionnaire and each is scored from 0( not at all) to 4(very much), for a maximum score of 48, higher score indicating lower financial toxicity.
financial toxicity experienced by patients as assessed by the COST - FACIT survey | 6 months after discharge
  This is a 12 item questionnaire and each is scored from 0( not at all) to 4(very much), for a maximum score of 48, higher score indicating lower financial toxicity.
financial toxicity experienced by patients as assessed by the COmprehensive Score for financial Toxicity (COST)-Functional Assessment of Chronic Illness Therapy (FACIT) survey | 12 months after discharge
  This is a 12 item questionnaire and each is scored from 0( not at all) to 4(very much). Questions 2,3,6 and 7 are reverse scored for a maximum score of 48, higher score indicating lower financial toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jonah Stulberg, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No